CLINICAL TRIAL: NCT06000540
Title: A Prospective Pilot Study to Evaluate the Safety, Tolerability and Efficacy of Utilizing Precise Computer Controlled Gas Challenge in Healthy Subjects for Identification of Coronary Artery Disease
Brief Title: Needle Free Assessment of Myocardial Oxygenation in Healthy Subjects
Acronym: NIMO-Healthy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15803
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Hypercapnia Group A (Experimental): Healthy subjects without a history of coronary artery disease will undergo computer-controlled gas challenges.
  Interventions: Device: RespirAct
- Hypercapnia Group B (Experimental): Healthy subjects without a history of coronary artery disease will undergo computer-controlled gas challenges.
  Interventions: Device: RespirAct
- Hypercapnia Group C (Experimental): Healthy subjects without a history of coronary artery disease will undergo computer-controlled gas challenges.
  Interventions: Device: RespirAct
- Hypoxia Group (Experimental): Healthy subjects without a history of coronary artery disease will undergo computer-controlled gas challenges.
  Interventions: Device: RespirAct

INTERVENTIONS:
Device: RespirAct — RespirAct device-based computer-controlled gas delivery at different concentrations as per protocol

SUMMARY:
This is a prospective pilot study to evaluate the safety, tolerability and efficacy of utilizing precise computer controlled gas challenge in healthy subjects for identification of coronary artery disease.

DETAILED DESCRIPTION:
This study will establish the safe and tolerable level of high PC02 and low P02 for future studies as potential stressors for coronary artery disease assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 45 years of age
2. No known cardiac disease

Exclusion Criteria:

1. Low blood pressure (systolic blood pressure < 100 mmHg)
2. Inability to voluntarily increase their breathing rate if prompted to do so
3. Persons with the inability to lie supine for 30-40 minutes
4. Persons who are pregnant, nursing, or implanted with intrauterine devices (IUD's)
5. Persons with significant neurological, pulmonary, renal or hepatic disease
6. Persons who have an abnormal cardiac rhythm or resting heart rate >100/min
7. Inability or unwillingness to provide informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Physiological Parameters Monitoring | 3 hours
  1. Saturation of peripheral oxygen as percentage
  2. Heart rate as beats per minute
  3. Noninvasive blood pressure as mmHg
  4. Partial pressure of oxygen as mmHg
  5. Partial pressure of carbon dioxide as mmHg
Assessment of Symptom Severity and Incidence | 3 hours
  1. Chest pain
  2. Headache
  3. Dizziness
  4. Confusion
  5. Fatigue
  6. Upset stomach
  7. Nausea
  8. Vomiting

SECONDARY OUTCOMES:
Participant Completion | Day 1 and Day 2
  Procedure tolerability will be evaluated by the number of participants completing day 1 and day 2 of study participation.
Patient comfort level score | 3 hours
  Participants will be asked to rate their comfort level for breathing from the mask and the gas changes as Painful, Not Comfortable, Tolerable for short time, tolerable for entire study, or comfortable.
Quality of Cardiac MRI | 3 hours
  The cardiac MRI images will be assessed for quality.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang HJ, Dey D, Sykes J, Butler J, Biernaski H, Kovacs M, Bi X, Sharif B, Cokic I, Tang R, Slomka P, Prato FS, Dharmakumar R. Heart Rate-Independent 3D Myocardial Blood Oxygen Level-Dependent MRI at 3.0 T with Simultaneous 13N-Ammonia PET Validation. Radiology. 2020 Apr;295(1):82-93. doi: 10.1148/radiol.2020191456. Epub 2020 Feb 25. PMID 32096705
- [Result] Poublanc J, Sobczyk O, Shafi R, Sayin ES, Schulman J, Duffin J, Uludag K, Wood JC, Vu C, Dharmakumar R, Fisher JA, Mikulis DJ. Perfusion MRI using endogenous deoxyhemoglobin as a contrast agent: Preliminary data. Magn Reson Med. 2021 Dec;86(6):3012-3021. doi: 10.1002/mrm.28974. Epub 2021 Oct 22. PMID 34687064
- [Result] Spano VR, Mandell DM, Poublanc J, Sam K, Battisti-Charbonney A, Pucci O, Han JS, Crawley AP, Fisher JA, Mikulis DJ. CO2 blood oxygen level-dependent MR mapping of cerebrovascular reserve in a clinical population: safety, tolerability, and technical feasibility. Radiology. 2013 Feb;266(2):592-8. doi: 10.1148/radiol.12112795. Epub 2012 Nov 30. PMID 23204541